CLINICAL TRIAL: NCT05034484
Title: A Randomized, Double-Blind, Placebo-Controlled Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of ALPN-303 in Adult Healthy Volunteers
Brief Title: A Study of ALPN-303 in Adult Healthy Volunteers
Acronym: RUBY-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alpine Immune Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AIS-D01
Record Dates: First submitted 2021-08-26; First posted 2021-09-05 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteer; BAFF; APRIL

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ALPN-303 Regimen A (Experimental)
  Interventions: Drug: ALPN-303
- Placebo Regimen A (Placebo Comparator)
  Interventions: Drug: Placebo
- ALPN-303 Regimen B (Experimental)
  Interventions: Drug: ALPN-303
- Placebo Regimen B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALPN-303 — Multiple dose levels will be evaluated.
  Arms: ALPN-303 Regimen A; ALPN-303 Regimen B
Drug: Placebo — Placebo will be administered
  Arms: Placebo Regimen A; Placebo Regimen B

SUMMARY:
This study is to assess the safety, tolerability, pharmacokinetics (the amount of drug in the blood), pharmacodynamics (how the drug effects the body) and immunogenicity (how the drug effects the immune system) of a single dose of an investigational drug called ALPN-303. Multiple dose levels will be tested.

ELIGIBILITY:
Summary of Inclusion Criteria:

* Able and willing to provide written informed consent
* Body mass index 18 to 32 kg/m2
* Agree to avoid strenuous physical activity for 2 days prior to each study visit
* Agree to use highly effective contraception during the study (all participants) and for 90 days after study drug dosing (males) or for 60 days after study drug dosing (females)
* Male participants must refrain from donating sperm during the study and for 90 days after study drug dosing
* Female participants must not be pregnant or breastfeeding and must refrain from donating ova during the study and for 60 days after study drug dosing
* Must have completed vaccination against SARS-CoV-2 at least 4 weeks prior to study drug dosing

Summary of Exclusion Criteria:

* Any current disease, condition, or treatment that could interfere with the study, interfere with interpretation of the data, or pose an unacceptable risk to the participant
* History or symptoms of significant psychiatric disease; mild, resolved depression or anxiety is acceptable
* History of immunological disorders, auto-immune disorders, acquired or congenital immune deficiency; see protocol for clarifications/exceptions
* History of significant hepatic or renal disease or impairment
* Evidence of an active or suspected cancer or a history of malignancy within the previous 3 years; see protocol for exceptions
* History of major organ transplantation with an existing functional graft
* Use or receipt of prescription medications, over-the-counter medications, herbal remedies, or investigation products (study drugs) within protocol-defined timeframes prior to study entry; hormone replacement therapy initiated at least 2 months prior to Screening is acceptable
* Significant loss of blood or blood product (including donation) over 500 mL or transfusion of any blood product during Screening or within 3 months of Screening
* Unwilling to refrain from alcohol use ≥ 48 hours prior to Study Day -1.
* Known hypersensitivity, allergy, or intolerance to ALPN-303, Fc-based biologic therapy, or any of the excipients contained in the ALPN-303 formulation
* Immunization with any live vaccine within 6 weeks prior to study drug administration, or expected to require any live vaccines during the study or within 6 weeks after receiving study drug
* Acceptable laboratory assessments at Screening and Day -1
* Positive screen for drugs of abuse or alcohol at Screening or Day -1
* Positive tests for infectious disease (HIV, hepatitis B, hepatitis C, SARS-CoV-2)
* Acute infection during or within 4 weeks prior to Screening
* History of frequent or atypical infections as defined per protocol; signs or symptoms of immunodeficiency
* History or presence of any chronic infectious condition
* Cardiac risk factors, as defined per protocol

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2021-11-15 (Actual); Primary Completion 2023-02-27 (Actual); Study Completion 2023-02-27 (Actual)

PRIMARY OUTCOMES:
Treatment-emergent Adverse Events (TEAE) | Day 1 through Day 30
  Type, incidence, and severity of TEAE as assessed by CTCAE

CONTACTS AND LOCATIONS:
Overall Officials: Stanford Peng, MD PhD, Study Director — Alpine Immune Sciences, Inc.
Locations (2):
- Australia (2):
  - Investigative Site, Brisbane, Queensland
  - Investigative Site, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No